CLINICAL TRIAL: NCT06183073
Title: Analgesic Efficacy of Transversus Abdominis Plane Block Versus Caudal Dexmedetomidine in Children Undergoing Abdominal Surgeries
Brief Title: Caudal Block With Bupivacaine and Dexmedetomidine Versus TAP Block With Bupivacaine Alone for Postoperative Analgesia in Pediatric Undergoing Infraumbical Surgeries
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Fouad Soliman, Lecturer of Anesthesia and ICU, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 2009
Record Dates: First submitted 2023-12-13; First posted 2023-12-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caudal block with bupivacaine and dexmedetomidine (Active Comparator): Caudal block with bupivacaine 0.25% in a dose of (1 ml / kg) and dexmedetomidine 1μg/ kg.
  Interventions: Procedure: caudal block; Drug: Dexmedetomidine; Drug: Bupivacain
- TAP block with bupivacaine (Active Comparator): TAP block with bupivacaine 0.25% in a dose of (0.5 ml / kg).
  Interventions: Procedure: TAP; Drug: Bupivacain

INTERVENTIONS:
Procedure: caudal block — bupivacaine 0.25% in a dose of (1 ml / kg)
  Other Names: bupivacaine
  Arms: Caudal block with bupivacaine and dexmedetomidine
Drug: Dexmedetomidine — dexmedetomidine 1μg/ kg.
  Arms: Caudal block with bupivacaine and dexmedetomidine
Procedure: TAP — analgesia
  Arms: TAP block with bupivacaine
Drug: Bupivacain — bupivacaine 0.25% in a dose of (0.5 ml / kg

SUMMARY:
Acute pain management for pediatric surgical patients intraoperatively and postoperatively is important for their comfort and psychological impact. Children aged 3-9 years old are included in the study and are divided randomly into two groups (45 children in each):

Group D: Caudal block with bupivacaine 0.25% in a dose of (1 ml / kg) and dexmedetomidine 1μg/ kg.

Group T: TAP block with bupivacaine 0.25% in a dose of (0.5 ml / kg).

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3-9 years old
* Physical status I and II class of the American Society of Anesthesiologists (ASA)
* Unilateral elective surgeries below the umbilicus

Exclusion Criteria:

* Parents or legal guardian refusal.
* History of developmental delay or mental retardation
* Contraindications to regional anesthesia as known or suspected coagulopathy, a known allergy to any of the study drugs, signs of infection at the site of caudal block.
* Hemodynamic unstable patient.

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2023-04-02 (Actual); Primary Completion 2024-01-14 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
1st analgesic requirement | 12 hours
  Time for first analgesic request (paracetamol intravenously 15 mg/kg) (h)

SECONDARY OUTCOMES:
Heart rate (HR) | 12 hours
  Hemodynamic assessment
systolic Blood Pressure (BP) | 12 hours
  Hemodynamic assessment
diastolic Blood Pressure (BP) | 12 hours
  Hemodynamic assessment
SpO2 -Hemodynamic assessment | 12 hours
Total paracetamol consumption | 12 hours
post operative pain score | 12 hours
  post operative pain score upon arrival to recovery room and then 2, 4,6, 8 , and 12 hours after surgery using Faces pain scale-revised.

CONTACTS AND LOCATIONS:
Overall Officials: Fouad I Soliman, MD, Principal Investigator — Sohag University
Locations (1):
- Fouad Ibrahim Soliman, Sohag, Egypt